CLINICAL TRIAL: NCT01104038
Title: EXCEL: Change in Cardiometabolic Disease Risk Factors During an Interactive Fitness Program
Acronym: EXCEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Laura Hayman, Associate Vice-Provost for Research & Professor of Nursing, University of Massachusetts, Boston
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: UMBCHB007; UL1RR025758-02 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Disease
Keywords: physical activity; cardiometabolic risk; children
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition Education/Lifestyle Counseling (Active Comparator): Children in this group will receive weekly group nutrition sessions , 30 minutes per week for 12 weeks, identical to those provided for the EXCEL intervention group and delivered by a registered dietician.
  Interventions: Behavioral: Nutrition Education ONLY
- EXCEL (Experimental): The EXCEL arm is the experimental arm of the study. Participants in this arm will receive supervised physical activity in the form of novel gaming (technology-mediated physical activity, 60 minutes per session, three times per week , for 12 weeks and 12 weeks of group nutrition education sessions.
  Interventions: Behavioral: EXCEL

INTERVENTIONS:
Behavioral: EXCEL — Children in the EXCEL intervention will receive 12 weeks of supervised physical activity, guided by principles of behavior change, in the form of exergaming (technology-mediated interactive physical activity)3 times per week for 12 weeks and will also receive weekly group nutrition education sessions
  Arms: EXCEL
Behavioral: EXCEL — Participants in the EXCEL intervention will receive 12 weeks of supervised physical activity in the form of exergaming (technology-mediated physical activity). Sessions will be held 3 times per week with 60 minutes of supervised physical activity.
  Other Names: EXERGAMING
  Arms: EXCEL
Behavioral: Nutrition Education ONLY — Children in the nutrition education group will receive 30 minutes per week of group nutrition education in the school environment and delivered by a registered dietitian The nutrition education sessions will be identical to those provided for the EXCEL group.
  Arms: Nutrition Education/Lifestyle Counseling

SUMMARY:
Childhood obesity has increased in prevalence over the past several decades and is predictive of adult type 2 diabetes and cardiovascular disease (CVD). Recent studies of children and youth suggest that exercise reduces cardiometabolic risk factors. Minimal data are available, however, on the effects of "exergaming" , interactive technology- mediated approaches to increasing physical activity in children and youth. This project involves a partnership between UMass Boston/GoKids Boston and Children's Hospital Boston featuring an interdisciplinary team of researchers and clinicians from pediatric cardiology, nursing, prevention and behavioral sciences and exercise physiology and is designed to examine the effects of exergaming on moderate or vigorous physical activity (MVPA) indices of adiposity, risk factors for cardiometabolic disease and self-competence in Boston Public School children. It is hypothesized that participation in the EXCEL/exergaming intervention for 60 minutes, three times per week for 12 weeks will significantly increase MVPA (as measured by accelerometers), pre- to- post intervention and compared to an Advice only (Nutrition Education) group.Results of this pilot study will guide and inform a larger study of exergaming in children from the Boston Public Schools.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grades 3-5
* able to attend GoKids and school-based weekly educational sessions for 12 weeks and complete baseline and follow-up testing
* informed consent from a parent or legal guardian and written assent from the child
* English speaking child
* free from medical conditions that would prohibit exercise as indicated by permission to participate in school physical education, and by review of screening questions with clearance from primary care provider as necessary.

Exclusion Criteria:

* abnormalities on screening/baseline evaluation that could pose a significant risk for exercise
* illness that would limit participation
* plans to move out of the area or change schools in the next 6 months

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change in moderate or vigorous physical activity (MVPA) between baseline and final visit (12 weeks) in children in the Excel intervention group as compared to children in the Advice only (Nutrition Education) group. | 12 weeks; follow up at 18 weeks
  The primary test of hypothesis is the comparison of change in MVPA between baseline and final visit (12 weeks) in children in the Excel intervention group as compared to children in the Advice-only (Nutrition Education) group. Accelerometers will be used to measure MVPA.

SECONDARY OUTCOMES:
pre-post EXCEL intervention changes in cardiorespiratory fitness and cardiometabolic risk factors (blood lipids, blood pressure, body mass index [BMI], waist circumference) | 12 weeks; follow-up at 18 weeks
  Cardiorespiratory fitness and cardiometabolic risk factors will be assessed at baseline and 12 and 18 weeks post-intervention in EXCEL intervention group and in the Advice only (Nutrition Education) group. Between and within group changes in cardiorespiratory fitness and cardiometabolic risk factors will be examined and compared at the 12 week and 18 week data point.

REFERENCES:
- [Derived] Crouter SE, de Ferranti SD, Whiteley J, Steltz SK, Osganian SK, Feldman HA, Hayman LL. Effect on Physical Activity of a Randomized Afterschool Intervention for Inner City Children in 3rd to 5th Grade. PLoS One. 2015 Oct 28;10(10):e0141584. doi: 10.1371/journal.pone.0141584. eCollection 2015. PMID 26510013